CLINICAL TRIAL: NCT01000545
Title: The Efficacy and Safety of Sulodexide in Filipino Diabetic Patients With Chronic Kidney Disease: A Randomized Controlled Trial
Brief Title: The Efficacy and Safety Study of Sulodexide in Filipino Diabetic Patients With Chronic Kidney Disease
Acronym: DEFINE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Corbridge Group Philippines, Inc. (Other)
Collaborators: Alfasigma S.p.A. (Industry)
Responsible Party: Mr. German A. Panghulan, Corbridge Group Philippines, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLD-CKD-001
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Kidney Disease
Keywords: Diabetes Mellitus; Chronic Kidney Disease; Glycosaminoglycans; Sulodexide; Macroalbuminuria; Safety and Efficacy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus | interventions — glucuronyl glucosamine glycan sulfate; Glycosaminoglycans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo gelcaps + best medical treatment (Placebo Comparator): Patient will receive 4 placebo gelcaps twice a day. Best Medical Treatment (BMT)refers to the treatment currently acceptable and standard measures for the decrease in proteinuria. These are strict blood sugar control (HBA1c < 7.0%) and BP control (BP< 130/80)
  Interventions: Drug: placebo capsules
- SLX 500LRU/day + best medical treatment (Active Comparator): Patient will receive 1 SLX gelcap and 3 placebo gelcaps twice a day.Best Medical Treatment (BMT)refers to the treatment currently acceptable and standard measures for the decrease in proteinuria. These are strict blood sugar control (HBA1c < 7.0%) and BP control (BP< 130/80)
  Interventions: Drug: Sulodexide
- SLX 1000LRU/day + best medical treatment (Active Comparator): Patient will receive 2 SLX gelcaps and 2 placebo gelcaps twice a day. Best Medical Treatment (BMT)refers to the treatment currently acceptable and standard measures for the decrease in proteinuria. These are strict blood sugar control (HBA1c < 7.0%) and BP control (BP< 130/80)
  Interventions: Drug: Sulodexide
- SLX 2000LRU/day + best medical treatment (Active Comparator): Patient will receive 4 SLX gelcaps twice a day. Best Medical Treatment (BMT)refers to the treatment currently acceptable and standard measures for the decrease in proteinuria. These are strict blood sugar control (HBA1c < 7.0%) and BP control (BP< 130/80)
  Interventions: Drug: Sulodexide

INTERVENTIONS:
Drug: Sulodexide — SLX 500 LRU, SLX 1000 LRU, SLX 2000 LRU per day to be taken orally for 12 months.
  Other Names: Vessel Due-F; SLX; Glycosaminoglycans
  Arms: SLX 1000LRU/day + best medical treatment; SLX 2000LRU/day + best medical treatment; SLX 500LRU/day + best medical treatment
Drug: placebo capsules — 8 soft-gel capsules per day to be taken orally for 12 months
  Other Names: placebo; placebo gelcaps
  Arms: placebo gelcaps + best medical treatment

SUMMARY:
The purpose of this study is to determine the effect and safety of Sulodexide in Filipino patients with Chronic Kidney Disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* positive 2 of 3 ACR > 300 mg/g or 24h urine protein or albumin collection > 300 mg/d in the absence of urinary tract infection
* serum creatinine 1.3 - 3 mg/dl in women and 1.5 - 3 mg/dl in men

Exclusion Criteria:

* age of onset of DM \< 18 years
* + renal disease like non-DM renal disease
* + CV diseases such as UA, MI, CABG
* + CVA or TIA within last 6 months
* untreated UTI

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1508 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-01 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
macroalbuminuria and serum creatinine | 52 weeks

SECONDARY OUTCOMES:
adverse events | 52 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- Philippines (7):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - Rizal Private Clinics, Metro Manila, Rizal
  - Holy Child Hospital, Dumaguete
  - Victoriano R. Potenciano Medical Center, Mandaluyong
  - Metropolitan Medical Center, Manila
  - Manila Adventist Medical Center, Pasay
  - The Medical City, Pasig